CLINICAL TRIAL: NCT04878861
Title: Rehabilitating Visual Deficits Caused by Stroke: Neurochemical and Neurophysiological Markers for Optimal Recovery
Brief Title: Rehabilitating Visual Deficits Caused by Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Rochester (Other); University of Turin, Italy (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, DrHollyBridge, Professor, University of Oxford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R60132/RE001
Record Dates: First submitted 2021-04-28; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Hemianopia; Hemianopsia; Quadrantanopia; Stroke Induced Vision Loss
Keywords: Vision; Stroke; Visual training; Blindsight; Visual pathway
MeSH Terms: conditions — Hemianopsia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Training in blind field (Experimental): All participants undergo this intervention. Internal control is comparing sighted and non-sighted parts of the field.
  Interventions: Behavioral: Training in the blind field

INTERVENTIONS:
Behavioral: Training in the blind field — Participants will complete visual training at two locations in the blind field. These two locations of training will be determined at the baseline study visit (0 months) and will be located within the perimetry-defined blind field. The training programme involves discriminating the direction of motion in a small circle of moving dots. The computer software and a chin-rest will be loaned to each participant to complete training at home. Participants will perform 300 trials at each location in their blind field, 5 days a week for at least 24 weeks (40-60 minutes in total). The computer programme will automatically generate a record of participant performance after each home training session.

SUMMARY:
This research aims to understand the efficacy of a visual training task to improve visual loss after stroke, also known as hemianopia. The investigators aim to understand whether training can improve vision and which areas or pathways in the brain are responsible for this improvement.

DETAILED DESCRIPTION:
Damage to the primary visual cortex (V1) due to stroke usually results in loss of visual function in half of the visual world, this is known as hemianopia. This visual loss can negatively affect quality of life, as most stroke survivors are no longer permitted to drive and have difficulties with navigation and socialising. There are currently limited treatment options, although recent evidence suggests that visual training can be effective in improving visual function (Huxlin et al, 2009; Cavanaugh & Huxlin, 2017). The aim of this research is to determine the capacity for visual rehabilitation after stroke using visual training and to understand the underlying brain mechanisms that might drive these improvements. This study will help the investigators to understand the brain mechanisms involved in visual rehabilitation and may allow the investigators to predict those most likely to benefit from visual rehabilitation in the future.

Twenty stroke survivors with hemi- or quadrantanopia will complete a 6-month visual motion discrimination training programme at home. Each participant will have three study visits; at baseline, 6-months and 9-months. At each visit the investigators will take measures of 1) visual fields 2) detailed tests of visual function 3) quality of life and 4) MRI scans of brain structure, function and neurochemistry. Between the baseline (0 month) and 6-month post-training session, participants will complete visual training at home. Between the 6-month post-training session and 9-month follow up, participants will not complete visual training at home. This study will therefore allow the investigators to determine whether rehabilitation improves conscious visual perception and quality of life as well as providing understanding of the neural mechanisms that underlie this improvement. The investigators will also determine whether improvements or neural changes persist after 3-months without training.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80
* Participant is willing and able to give informed consent for participation in the study
* Fluent English-speaking healthy adults
* Has suffered damage to the visual cortex at least 6 months before the study

Exclusion Criteria:

* Previous eye disease or impairment other than hemianopia
* Neurological or psychiatric illness
* Contraindication to MRI
* Pregnant or breast feeding
* Second stroke during training

Data quality assurance (participant data will be removed from analysis for the following reasons):

* Concurrent participation in other "vision therapy"
* Unreliable visual fields, indicated by greater than 20% fixation losses, false positives, or false negatives
* Inability to demonstrate fixation stability on eye movement monitored testing
* Failure to complete at least 100 training sessions over 6-months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-13 (Actual); Primary Completion 2024-10-16 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Change in motion discrimination thresholds after 6 months of training | 6 months
  Change in normalised discrimination thresholds on psychophysical motion discrimination task at two trained locations between baseline (0-month) and 6-month follow up. These assessments will be based on what motion can be reliably detected at a 75% correct level of performance.

SECONDARY OUTCOMES:
Maintenance of improvement in motion discrimination thresholds at 9-month follow up. | 9 months
  No change in normalised discrimination thresholds on psychophysical motion discrimination task at two trained locations between 6-month and 9-month follow up. These assessments will be based on what motion can be reliably detected at a 75% correct level of performance.
Change in area improved on the Humphrey perimetry (24-2 and 10-2) | 6 months
  Change in area improved on a composite measure of deficit size calculated from 24-2 and 10-2 across both eyes. Area of improvement will be calculated as the area where the sensitivity improved by more than 6 decibels (dB) relative to pre-training.
Maintenance area improved on the Humphrey perimetry (24-2 and 10-2) | 9 months
  No change in area improved on a composite measure of deficit size calculated from 24-2 and 10-2 across both eyes. Area of improvement will be calculated as the area where the sensitivity improved by more than 6dB relative to pre-training.
Change in contrast detection at trained locations | 6 months
  Change in detection of stimulus at 1%, 5%, 10%, 50% and 100% contrast baseline (0-month) and 6-month follow up.
Maintenance contrast detection at trained locations | 9 months
  No change in detection of stimulus at 1%, 5%, 10%, 50% and 100% contrast between the 6-month and 9-month follow up.
Change in visual quality of life | 6 months
  Change on the Visual Function Questionnaire 25 between baseline (0-month) and 6-month follow up.
Maintenance of visual quality of life | 9 months
  No change in visual quality of life as measured by the Visual Function Questionnaire 25 between 6-month and 9-month follow up.
Change in white matter integrity | 6 months
  Change in white matter integrity in lateral geniculate nucleus (LGN) to extrastriate motion area (hMT+) and LGN to primary visual cortex (V1) tracts between baseline (0-month) and 6-month follow up, assessed by diffusion-weighted imaging
Maintenance of white matter integrity | 9 months
  No change of integrity in LGN-hMT+ and LGN-V1 tracts between 6-month and 9-month follow up, assessed by diffusion-weighted imaging.
Change in neurochemistry | 6 months
  Change in neurochemistry in visual motion area, hMT+ between baseline (0-month) and 6-month follow up, assessed by Magnetic Resonance Spectroscopy (MRS).
Maintenance of neurochemistry | 9 months
  No change in neurochemistry in visual motion area, hMT+ between 6-month and 9-month follow up, assessed by Magnetic Resonance Spectroscopy (MRS).
Change in brain activity during visual stimulation (Blood-oxygen-level-dependent imaging, or BOLD, signal change) | 6 months
  Change in brain activity during moving visual stimulation, assessed by functional magnetic resonance imaging (BOLD signal) in visual motion area, hMT+ between baseline (0 month) and 6-month follow up.
Maintenance of brain activity during visual stimulation (BOLD signal change) | 9 months
  Maintenance of brain activity during moving visual stimulation, assessed by functional magnetic resonance imaging (BOLD signal) in visual motion area, hMT+ between the 6-month and 9-month follow up.
Change in resting state connectivity | 6 months
  Change in resting state connectivity in the visual cortex between baseline (0-months) and 6-months, assessed by resting state functional magnetic resonance imaging (BOLD signal)
Maintenance of resting state connectivity | 9 months
  Maintenance of resting state connectivity in the visual cortex between 6-month and 9-month follow up, assessed by resting state functional magnetic resonance imaging (BOLD signal)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Bridge, PhD, Principal Investigator — University of Oxford
Locations (1):
- Wellcome Centre For Integrative Neuroimaging, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to share subsets of the data as appropriate.
Time Frame: After conclusion of study.